CLINICAL TRIAL: NCT03730831
Title: Childhood Maltreatment, Traumatic Experiences and Stress-associated Parameters: Relationship and Influence on the Course of Illness in Schizophrenia Spectrum Disorders
Brief Title: Childhood Maltreatment, Traumatic Experiences and Stress-associated Parameters in Schizophrenia Spectrum Disorders
Acronym: NETPSYCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Konstanz (Other)
Collaborators: Centre for Psychiatry Reichenau (Unknown)
Responsible Party: Principal Investigator, Michael Odenwald, Head of psychological outpatient clinic, head of psychology at the research ward, University of Konstanz
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NET PSYCH 2018
Record Dates: First submitted 2018-07-05; First posted 2018-11-05 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Schizophrenia Spectrum Disorder; PTSD
Keywords: Course; Schizophrenia Spectrum Disorder; Posttraumatic Stress Disorder; Narrative Exposure Therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (second work program) (Experimental): Narrative Exposure Therapy Narrative Exposure Therapy (NET) is a brief manualized trauma-focussed psychotherapeutic treatment and will be performed according to the manual of Schauer et al., 2011. In NET, traumatic experiences are worked through and placed in the context of the entire life story.
  Interventions: Behavioral: Narrative Exposure Therapy

INTERVENTIONS:
Behavioral: Narrative Exposure Therapy — 8-20 sessions: 1 lifeline session, 6-17 sessions narrative exposure, 1-2 sessions of future-oriented counselling
  -> Intervention is a part of the second work program. First work program focueses on cross-sectional data and includes a systematic record of psychopathology in participants with schizophrenia sepctrum disorder.

SUMMARY:
Childhood maltreatment (CM) in psychotic disorders is associated with increased cognitive deficits, severe psychotic symptoms, and increased comorbidity. The number of different stress experiences also increases the probability of trauma-associated symptoms. Furthermore, neurobiological changes play a key role in the vulnerability of individuals with early traumas for mental and physical illnesses, among others for diseases of the schizophrenia spectrum disorder and the further course of the disease.

The project is divided into two work programs and pursues:

1. A detailed recording of the course of symptoms in participants with schizophrenia spectrum disorder to link this data with a systematic recording of CM and traumatic experiences and biological data.
2. On a subsample of participants with schizophrenia spectrum disorder and a comorbid post-traumatic stress disorder (PTSD), the researchers want to investigate whether symptom traits of existing psychotic disorders, trauma-associated symptoms and cognitive functions can be influenced by a trauma-specific treatment (NET), that has been proven to be effective in the treatment of PTSD.

DETAILED DESCRIPTION:
Numerous scientific findings point to the influence of CM and traumatic experiences on the risk of mental and physical illnesses, their severity and their course. Traumatic experiences also increase the risk of demonstrating psychotic symptoms or even develop psychotic disorders. Furthermore, the number of different stress experiences also increases the probability of trauma-associated symptoms (symptoms of post-traumatic stress disorder (PTSD) and dissociative experiences).

Neurobiological changes in the immune system, the defense of stress and also central nervous circuits and structures play a key role in the vulnerability of individuals with early traumas for mental and physical illnesses, e.g. for diseases of the schizophrenia spectrum disorder and the further course of the disease.

The recording of stressful and traumatic life experiences has been largely neglected in everyday clinical practice, especially in patients with a schizophrenia spectrum disorder. The diagnosis of PTSD is rarely given in everyday clinical practice, so that trauma-specific treatment is often not offered.

The targeted use of a scientifically proven intervention to reduce the symptoms of PTSD (NET: Narrative Exposure Therapy) involves a change in stress-associated biomolecular parameters and normalizes neuronal brain activity.

The project pursues a systematic assessment of CM and traumatic experiences as well as a detailed recording of the course of symptoms in participants with schizophrenia spectrum disorder. Furthermore, in a subsample of participants with schizophrenia spectrum disorder and comorbid PTSD, the researchers want to investigate whether symptom traits of existing psychotic disorders, trauma-associated parameters and cognitive functions can be influenced by a trauma-specific treatment (NET).

The original research plan had to be modified because of the COVID-19 restrictions. Thus, during the course of the study, we had to modify design and data assessment.

The original plans related to the two work programs of the study and their modification are described below:

Work program 1 (WP1):

Originally, the WP1 included a weekly prospective assessment of psychotic symptoms on a sample of n=100 participants with schizophrenia spectrum disorder and planed to link this data with results from a cross-sectional assessment on traumatic and childhood maltreatment and biological data (cortisol awakening (CAR), diurnal cortisol profile, tonic cortisol concentration in hair and determination of mitochondrial respiratory activity in mononuclear cells).

Modifications of the original study plan of WP1:

1. Originally, it was planned to examine the determination of mitochondrial respiratory activity in mononuclear cells. Due to a change in cooperation with a partner study project, examination of mitochondrial respiratory activity in mononuclear cells was later on excluded and focus was set only on the endocrine system via cortisol response (CAR, diurnal cortisol profiles and hair cortisol concentration).
2. Due to the COVID pandemic, saliva samples could only be collected before pandemic restriction rules. Therefore, not all participants contributed in all parts of the originally planned WP1.
3. Due to COVID restrictions, access to the study population was restricted and the planned total of n=100 could not be completed, instead n=79 patients could be included into the study.
4. In addition to the patient data, we also collected data from healthy controls (n=39) to replicate existing findings between healthy controls and people with schizophrenia spectrum disorder.
5. In addition to the clinical interview (cross-sectional assessment) of traumatic and childhood maltreatment, we included measurements of parental bonding (high/low parental care, high/low overprotection) to have a more detailed look on how childhood experiences can influence symptom course of psychotic disorders.
6. The weekly assessment of psychotic symptoms did not proof to be feasible in daily clinical routine due to the high time consumption of assessments during COVID restrictions. Outcome measures therefore focused on three points in time, i.e. admission to study, 4 weeks after admission, and 3 months after admission or - if released earlier - at release from inpatient treatment.

The adapted WP1 pursued the following research questions:

1. What influence do childhood maltreatment and traumatic experiences have on current psychological and physical well-being (systematic & detailed symptom recording)?
2. What influence does the family atmosphere have on the illness course?
3. Do parameters of the stress hormone system (wake-up cortisol, diurnal cortisol profile, hair cortisol concentration) correlate with measures of past childhood maltreatment, traumatic experiences, and parental bonding?

   Work program 2 (WP2):

   The second work program originally focussed on the subgroup of WP1 participants with schiziphrenia spectrum disorder and comorbid PTSD. It was planned to conduct a randomized controlled pilot study with n=20 to determine the impact of trauma-focused therapy (NET) on the course of symptoms. In addition to the symptoms of PTSD, psychosis-specific parameters such as cognitive functions and biological characteristics were planned to be repeatedly recorded (pre, post, 6 months and 12 months after completing trauma therapy).

   Modifications of the original study plan of WP2:
   1. Originally, a randomized control pilot study was planned with n=20 participants randomly allocated to either an active intervention group (n=10, receiving NET additionally to care as usual) or to a no treatment group (care as usual; n=10). Due to restricted manpower and lowered feasibility in clinical daily routine during COVID, our study design had to be adapted and the control group had to be omitted. In stead, we conducted a case series of the 10 cases who received the active treatment. The adapted study, therefore, had a single-group, pre-test, post-test, and follow-up-test design.
   2. We planned to implement 6-10 trauma therapy sessions of 90 minutes per case. Due to the specific nature of psychotic disorders (e.g., conceptual disorganization or limited cognitive capacities), the NET routine had to be adapted. For example, the length of the sessions often had to be shortened, which led in most cases to a higher number of sessions as planned (on average 15-20 sessions). For more details, see our publication: Breinlinger, S., Pütz, A.-K., Stevens, N. R., Mier, D., Schalinski, I., & Odenwald, M. (2020). Narrative Exposure Therapy in challenging cases and conditions. Maltrattamento e Abuso All'Infanzia: Rivista Interdisciplinare, 22(3), 37-50. https://doi.org/10.3280/MAL2020-003004.
   3. Furthermore, the follow-up assessment was changed to only pre (T0), post (T1) and 6 month follow-up (T2, 6 months after completing NET) for all measurements (PTSD symptoms, dissociation, cognitive functions, psychotic symptoms, depression, suicidal tendencies, quality of life).
   4. In the longitudibal course of WP2, biological data were only assessed at T1 (see reasons above relating to COVID pandemic). Instead, focus was set on clinical parameters: Primary outcomes were diagnosis, symptom severity of PTSD and dissociation assessed at T0, T1 and T2. Secondary outcomes were depressive symptoms, psychotic symptoms, suicidal tendencies, quality of life and cognitive performance measured by a standardized test battery. Single t-tests were used for data analysis.

   WP2 therefore pursued the following research questions:
4. What changes of trauma-related and psychotic symptoms can be observed in patients with schizophrenia spectrum disorder and PTSD after a specific PTSD treatment module?

Giving the division of the work program in a cross sectional and a prospective part, our original study title "Narrative Exposure Therapy in Patients With Psychotic Disorders and a Posttraumatic Stress Disorder" included only WP2. In order to place both work programs in an overall context, the overall title was changed to:

"Childhood maltreatment, traumatic experiences and stress-associated parameters: Relationship and influence on the course of illness in schizophrenia spectrum disorders."

ELIGIBILITY:
Inclusion Criteria for the first work program:

- Patients with schizophrenia spectrum disorder

Inclusion Criteria for the second work program:

- Patients with schizophrenia spectrum disorder and comorbid PTSD Diagnosis (DSM-5)

Exclusion Criteria (1st and 2nd work program):

* mental impairment (e.g. dementia)
* insufficient language comprehension
* non-compliance with appointments

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-10-24 (Actual); Study Completion 2022-10-24 (Actual)

PRIMARY OUTCOMES:
PTSD symptom severity (PCL-5) | 1st. work program: at baseline. 2nd work program: Change from baseline (T0) to post treatment (T1; 1 week after completing NET) and 6-month follow-up (T2, 6 months after completing NET)
  PTSD symptoms are measured in interview process (reporting period: previous 4 weeks) with the PTSD Checklist - 5 (PCL-5; Weathers, Litz, et al., 2013).
Psychotic Symptom Severity | 1st workprogram: Change from admission to 4 weeks and 3 months after admission or if earlier at release; 2nd workprogram: Change of psychotic symptoms from baseline (T0) to post (T1; 1 week after completingNET) and 6 months follow-up (T2)
  The course of psychotic symptoms is measured during inpatient treatment (from admission to study to release from inpatient treatment, typically for 6-8 weeks) with the Positive and Negative Syndrome Scale (PANSS; Kay, S. R., Fiszbein, A., & Opfer, L. A. (1987).
Dissociation (Shut-D) | 1st. work program: at baseline. 2nd work program: Change from baseline (T0) to post-treatment (T1; 1 week after completing NET) and 6 months follow-up (T2; 6 months after completing NET)
  Dissociative symptoms are assessed using the Shutdown Dissociation Scale (Shut-D), which measures the frequency of symptoms such as fainting, blurred vision, dizziness, altered hearing or vision, numbness, paralysis, and others {Schalinski, 2015 #46}. Participants reported the frequency of these symptoms over the past 6 months on a scale from 0 (not at all) to 3 (several times a week), with a total score ranging from 0 to 39.
Childhood maltreatment including parental bonding/family atmosphere | 1st and 2nd work program: at baseline.
  CM are assessed using the Maltreatment and Abuse Chronology of Exposure scale (MACE; {Teicher, 2015 #73}; German version KERF by {Isele, 2014 #44}) developed to retrospectively assess exposure to ten types of CM from infancy to age 18, encompassing abuse (such as physical, verbal, and non-verbal emotional abuse, witnessing interparental and sibling abuse, peer-related verbal abuse and physical bullying, and intra-, extra-familial, or peer-related sexual abuse) as well as emotional and physical neglect.
cortisol awakening response (CAR), diurnal cortisol profile and corresponding hair cortisol concentration | only 1st work program: CAR at awaking, 30, 45 and 60 minutes after awakening; at noon (directly before lunch) and in the evening (directly before dinner); Hair cortisol concentration once
  During the first hour after awakening saliva samples will be repeatedly collected following the established procedure.

SECONDARY OUTCOMES:
MATRICS Consensus Cognitive Battery | only 2nd work program: Change in cognitive functions is measured at baseline (T0), post-treatment (T1; within 1 month after completing NET) and 6 months follow-up (T2; 6 months after completing NET)
  Cognitive change is measures with the MATRICS Consensus Cognitive Battery (Nuechterlein et al., 2008)
Depression Severity | 1st. workprogram: at baseline. 2nd work program: Change in depression severity is measured at baseline (T0), post-treatment (T1; within 1 week after completing NET) and 6 months follow-up (T2; 6 months after completing NET)
  Changes in depressive symptoms measured with Beck DEpression Inventory revised (BDI-II)
Suicidal tendenies | 1st. workprogram: at baseline. 2nd work program: Change in suicidal tendencies is measured at baseline (T0), post-treatment (T1; within 1 week after completing NET) and 6 months follow-up (T2; 6 months after competing NET)
  MINI International Neuropsychiatric Interview (M.I.N.I.), Suicidal Scale (Lecrubier et al., 1997)
Changes in quality of life | 1st. workprogram: at baseline. 2nd work program: Change in quality of life is measured at baseline (T0), post-treatment (T1; within 1 week after completing NET) and 6 months follow-up (T2; 6 months after completing NET)
  WHO Disability Assessment Schedule (WHODAS 2.0; World Health Organization, 2010)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Konstanz, Psychotherapy Outpatient Clinic, Konstanz, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nuechterlein KH, Green MF, Kern RS, Baade LE, Barch DM, Cohen JD, Essock S, Fenton WS, Frese FJ 3rd, Gold JM, Goldberg T, Heaton RK, Keefe RS, Kraemer H, Mesholam-Gately R, Seidman LJ, Stover E, Weinberger DR, Young AS, Zalcman S, Marder SR. The MATRICS Consensus Cognitive Battery, part 1: test selection, reliability, and validity. Am J Psychiatry. 2008 Feb;165(2):203-13. doi: 10.1176/appi.ajp.2007.07010042. Epub 2008 Jan 2. PMID 18172019
- [Background] Kay SR, Fiszbein A, Opler LA. The positive and negative syndrome scale (PANSS) for schizophrenia. Schizophr Bull. 1987;13(2):261-76. doi: 10.1093/schbul/13.2.261. PMID 3616518